CLINICAL TRIAL: NCT04713774
Title: Evolution of Bone Density, Bone Micro-architecture and Vascular Calcifications in Patients After Kidney Transplantation
Brief Title: Bone Density and Vascular Calcifications Evolution After Renal Transplant
Status: Recruiting | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Antoine Bouquegneau, Principal Investigator, University of Liege
Other Study IDs: Liege REBON Vasc
Record Dates: First submitted 2021-01-08; First posted 2021-01-19 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Kidney Transplant; Complications; Bone Loss
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: High-resolution peripheral quantitative CT scanner (HRpQCT) — HR-pQCT images of the distal radius and distal tibia (non-dominant, non-fractured limb) will be obtained using the XtremeCT device with standard protocols. HR-pQCT images wil be analysed with standard software and extended cortical measures software. This software identifies the periosteal and endosteal boundaries, enabling assessment of cortical micro- structural bone properties, including apparent cortical thickness (Ct.Th, mm), cortical tissue mineral density (TMD, mgHA/cm3) and cortical porosity (Ct.Po, %).

SUMMARY:
The investigators project is based on:

* Assessment of bone architecture by high resolution peripheral scanner (HRpQCT) and bone densitometry (DEXA);
* The non-invasive detection of vascular calcifications (by abdominal CT scanner) and bone abnormalities associated with kidney transplantation, as well as the analysis of evolution over time;
* Longitudinal evaluation of nephrological clinical parameters (glomerular filtration rate, number and type of rejections, immunosuppressive medications) as well as biological and urinary parameters of mineral metabolism (parathormone, sclerostin, bone alkaline phosphatase) depending on the type and severity of bone abnormalities;
* The evaluation of these nephrological clinical parameters and of the biological parameters of mineral metabolism depending on the extent and evolution of vascular calcifications but also on bone morphology;
* The study of possible relationships between bone mass and muscle mass (and functioning)

DETAILED DESCRIPTION:
Bone and mineral abnormalities are frequent in kidney transplant patients and are associated with a high risk of fracture, cardiovascular mortality, but also with an increase in the frequency of hospitalisations and thus healthcare's costs. The pathophysiology of bone disorders appearing after transplantation arises from a complex interaction between different factors. These include both pre-transplant renal osteodystrophy lesions and bone loss associated with the kidney transplant itself. This bone loss results from a variety of causes. The management of these bone abnormalities is complex in daily clinical practice because only the bone biopsy can accurately determine the type of abnormality present, and this examination is rarely performed due to its invasive nature. The link between the development of bone abnormalities and the presence or even the progression of vascular calcifications remains very poorly understood. This link is however fundamental because vascular calcifications could explain the increased risk of cardiovascular mortality in these patients. Understanding and diagnosing bone abnormalities early, ideally in a non-invasive manner, could help prevent bone and vascular degradation frequently found after renal transplantation.

Despite significant improvement in recent years, mortality as well as cardiovascular morbidity remain very high in kidney transplant patients. The reported annual risk of fatal or non-fatal cardiovascular events is 3.5% to 5%, even after adjusting for traditional risk factors (such as diabetes, hypertension, obesity, smoking and dyslipidemia). Certain factors related to chronic kidney disease (CKD) or transplant appear to influence the high incidence of cardiovascular events. These include, among others, the duration of dialysis before the transplant, the function of the graft after transplantation, proteinuria, episodes of acute rejection, new cases of post-transplant diabetes, the toxic effects of immunosuppressive drugs but also the bone metabolism abnormalities observed in transplant patients.

It is therefore essential to be able to accurately assess the presence of abnormalities in bone metabolism by non-invasive techniques and thus to determine whether or not there is a link between them and cardiovascular morbidity and mortality. This allows appropriate management as well as a precise assessment of the impact of new drugs on bone metabolism and the future of transplant patients.

Currently, the clinical management of bone abnormalities includes the use of surrogate biochemical markers such as parathyroid hormone (PTH), bone alkaline phosphatases (bPhA), osteoprotegerin (OPG), the N-terminal propeptide of procollagen type I (P1NP), tartrate resistant acid phosphatase type 5b (TRAP5b), C-terminal collagen type I telopeptides (CTX), osteocalcin and sclerostin. There are conflicting data in the literature as to their correlation with histological and histomorphometric analysis of bone biopsies. These biomarkers tend to take a place in the diagnosis and in the follow-up of patients with abnormalities of bone metabolism, as well as possibly in the detection of vascular calcifications. However, the effectiveness and reliability of this biochemical approach remain to be demonstrated.

On the other hand, imaging techniques allow us to approach the bone structure. They could therefore also be associated with biomarkers to replace bone biopsy. Bone density by bi-photonic x-ray absorptiometry (DEXA) is a relatively accurate and non-invasive screening method for estimating bone mass, mainly trabecular, and which appears to help predict the risk of fracture in kidney transplant patients. DEXA is, however, unable to assess the microarchitecture of bone and only provides a two-dimensional assessment of bone density. The correlation between BMD and fracture risk is, however, much less clear in patients with renal impairment and some studies sometimes even find an absence of correlation. Currently a new software used in DEXA, the Trabecular Bone Score (TBS), seems to help in the assessment of bone microarchitecture. This score is most often weighted with the FRAX to give a better value of the fracture risk. Some data currently appear in the normal population, but no robust data are present in kidney transplant patients.

On the other hand, the peripheral high-resolution scanner (HRpQCT) provides information on the bone micro-architecture as well as a quantitative measurement of the volumetric density of the cortical bone, which is more impacted during renal failure, and. In this context, the investigators goal in this study is to collect all of these biological and imaging data in order to predict the underlying bone histomorphometry.

The analysis of bone density by DEXA will be carried out at the vertebral, hip and wrist level as a direct result of the transplantation (first 10 days post transplant) at 3 months and then annually for all renal transplant patients included in the study. Analysed of the relevance of this examination for the detection of BMD and long-term fracture risk (longitudinal study). The TBS will also be assessed by the same exam to assess its sensitivity for the detection of fracture risk.

The high-resolution scanner will be performed on the distal part of the radius and tibia for the evaluation of bone micro-architecture. This examination will be performed at the same frequency as the DEXA.

Then we will evaluate prospectively (at 3 months and 12 months) with a longitudinal follow-up the various BMD data related to the presence and evolution of vascular calcifications (see below) detected by DEXA as well as the various blood and urinary biomarkers.

Markers such as vitamin D, Ca2 +, PTH, bPhA, OPG, P1NP, TRAP5b, CTX, osteocalcin, sclerostin, vitamin K and the decarboxylated and dephosphorylated form of the matrix-Gla protein (MGP), and intact fibroblast growth factor 23 (FGF23) will be evaluated in order to seek a possible link with graft survival, the development of vascular calcifications and the risk of fractures. Depending on the results of the DEXA performed and if a therapeutic indication is considered in the context of fracture osteoporosis (bisphosphonates, denosumab), the patients will be followed prospectively and their data will be collected.

A measurement of DEXA and bone microarchitecture by HRpQCT will also be carried out bilaterally in the upper limbs in order to assess the impact of the location of the arteriovenous fistula on bone density in view of the possible impact described in the literature on a population of hemodialysis patients

The assessment of renal fibrosis will also be analyzed on the basis of renal biopsies performed routinely in transplant patients at 3 months and in the event of biopsies performed due to deterioration of renal function. The assessment of the degree of fibrosis will be analyzed in light of the abnormalities of the phosphocalcic balance to see if a link between the two exists.

Currently the reference technique for the detection of calcifications remains the chest scanner with detection of CAC. This tedious and irradiating technique is however difficult to use in current clinical practice. Calcifications of the abdominal aorta (AA) are as important as CAC and are associated with sudden death mortality in patients with renal failure. In the general population, the detection of calcifications by CT scan or by lateral radiography at the AAA level (AAB profile) has shown good correlations with the level of CAC. In the general population, the measurement of AA calcifications based on the lateral radiography images used during DEXA also seems to demonstrate good sensitivities and specificities, when the images obtained by DEXA are compared to the radiography of the AAB and to detection of AA calcifications by CT scan. In a population of transplant patients, the demonstration of calcifications via DEXA was associated with the risk of cardiovascular mortality of patients but has never been compared to the profile blank abdomen which remains the standard technique. In the population of kidney transplant patients, the literature has not established a link between the detection of calcifications by these two techniques (DEXA and abdominal scan) on the risk of cardiovascular events.

The hypothesis is that the detection and follow-up of calcifications in the aorta could only be done with this simple and rapid test, DEXA, and that it could therefore be combined with the measurement of BMD. We will therefore study the correlation between calcifications of the abdominal aorta detected by abdominal CT scan and those detected by DEXA.

The first objective is to prospectively study between 40 and 50 transplant patients. We will measure the calcifications observed by DEXA and follow them over time (first measurement carried out 3 months after transplant, and then once a year). Correlation analyzes will be performed to assess the sensitivity of the different techniques for the detection of calcifications both between techniques (abdominal CT scan during the first 10 days post-transplant and at 1 year) as well as between observers (3 observers: radiologist, nephrologist and rheumatologist). A measurement of the difference in calcifications according to the examinations will be evaluated to make it possible to assess the evolution of calcifications in the same patient according to the different clinical and biological parameters

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Recent kidney transplant patients (<3 months)
* Medical history available
* Biological parameters of the past year available

Exclusion Criteria:

* Treatment with bisphosphonate, RANKL inhibitor or SERM with bone action in the last 3 months before the transplant
* Multiple organ transplant patients

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Kidney recipients aged over 18 and of all sexes recruited from the Centre Hospitalier Universitaire de Liege
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-12-12 (Estimated); Study Completion 2026-12-13 (Estimated)

PRIMARY OUTCOMES:
Bone density evolution | At 1 year
  Evolution of bone density after kidney transplantation
Bone density evolution | At 2 year
  Evolution of bone density after kidney transplantation
Bone micro-architecture evolution | At 1 year
  Bone micro-architecture evolution evaluate by HRpQCT after kidney transplantation
Bone micro-architecture evolution | At 2 year
  Bone micro-architecture evolution evaluate by HRpQCT after kidney transplantation

SECONDARY OUTCOMES:
Vascular calcification evolution | At 1 year
  Evolution of vascular calcification evaluated by abdominal calcification score on CT-SCan after kidney transplantation
Vascular calcification evolution | At 3 months, 1 year and 2 years
  Evolution of vascular calcification evaluated by abdominal calcification score on CT-SCan after kidney transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Bouquegneau, Principal Investigator — University of Liege
Locations (1):
- Centre Hospitalier Universitaire de Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No